CLINICAL TRIAL: NCT03890744
Title: A Multicentre Phase IIa Study to Evaluate the Efficacy and Tolerability of ModraDoc006/r in Patients With Recurrent or Metastatic HER-2 Negative Breast Cancer, Suitable for Treatment With a Taxane
Brief Title: ModraDoc006/r in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Modra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18DMB
Record Dates: First submitted 2019-01-31; First posted 2019-03-26 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 14 evaluable patients will be treated in the first stage (Stage A) of this Simon two-stage minimax designed trial. If 0 or ≥ 2 objective responses at week 8 (with confirmation at week 12) are observed in Stage A, no further patients will be enrolled. If 1 objective response is observed, an additional 10 patients with recurrent or metastatic HER-2 negative breast cancer will be included in the second stage (Stage B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ModraDoc006/r (Experimental): Weekly ModraDoc006/r treatment as ModraDoc006 (oral docetaxel) 10mg tablets combined with ritonavir 100mg tablets
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — Treatment with twice daily once weekly (BIDW) ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets
  Other Names: oral docetaxel formulation

SUMMARY:
This is a multicenter phase IIa study to evaluate the efficacy and tolerability of ModraDoc006 in combination with ritonavir (denoted ModraDoc006/r) in patients with recurrent or metastatic HER-2 negative breast cancer, that are suitable for treatment with a taxane as 1st-3rd line of therapy.

DETAILED DESCRIPTION:
This is a phase IIa, multicentre, two-stage, single-arm, clinical study with the primary objective is to determine the efficacy of ModraDoc006 in combination with ritonavir (denoted ModraDoc006/r) in patients with recurrent or metastatic HER-2 negative breast cancer, as measured by RECIST v1.1 criteria of objective response rate (ORR). To this aim, a Simon two-stage minimax design will be used, in which 14 evaluable patients will be treated in the first stage (Stage A). If 0 or ≥ 2 objective responses at week 8 (with confirmation at week 12) are observed in Stage A, no further patients will be enrolled. If 1 objective response is observed, an additional 10 patients with recurrent or metastatic HER-2 negative breast cancer will be included in the second stage (Stage B).

All patients will be treated with ModraDoc006/r, given as oral tablets twice daily once weekly (BIDW).

Patients will be radiologically assessed at week 8 and 12 by CT scan (or MRI if CT is contraindicated), and may continue to receive study medication with ongoing radiological scans every 6 weeks until disease progression (according to RECIST v1.1), unacceptable toxicity, or discontinuation for any other reason.

Furthermore, the safety and tolerability of ModraDoc006/r in the target population will be assessed. Additionally, as metastatic breast cancer may occur at older age, often coinciding with other non-malignant diseases and co-medications, this protocol investigates whether ModraDoc006/r can be applied safely in these (frail) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and to comply with the protocol
2. Histologically- or cytologically confirmed diagnosis of recurrent or metastatic HER-2 negative breast cancer
3. Female of age 18 years or above
4. Patients who are eligible to receive a taxane as monotherapy as 1st-3rd line of therapy for recurrent or metastatic breast cancer. A maximum of two previous lines of chemotherapy is allowed (including experimental i.e. non-registered chemotherapy alone or in combination). Re-treatment with one of the same drugs after treatment interruption for reasons of patient preference and/or progression of disease counts as a new treatment
5. WHO performance status of 0, 1 or 2 (Appendix II)
6. Estimated life expectancy of at least 12 weeks
7. Resolution of toxicity of prior therapy to < grade 2 (except for alopecia and transaminases in case of liver metastases) as defined by CTCAE v5.0 (Appendix III)
8. Evidence of measurable disease present at baseline as defined by RECIST v1.1
9. Able and willing to swallow oral medication
10. Able and willing to undergo radiologic scans (CT scan, or MRI if CT is contraindicated)
11. All patients of childbearing potential must have a negative high sensitive pregnancy test at screening (urine/serum) and agree to use highly effective method for contraception from time of signing Informed Consent until at least 12 weeks after the last administration of study drug
12. Laboratory criteria:

    * Platelet count ≥ 100 x 109 /L
    * Haemoglobin ≥ 6.0 mmol/L or 9.67 g/dL
    * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109 /L
    * Total bilirubin ≤ 1.5 x ULN, except for patients with familial bilirubinaemia (Gilbert's disease)
    * Serum ASAT and ALAT ≤ 2.5 x ULN (≤ 5 x ULN with liver metastases)
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula or MDRD [Modification of Diet in Renal Disease])

Exclusion Criteria:

1. Systemic chemotherapy or radiation therapy within the last 4 weeks, endocrine based therapy and CDK4/6 inhibitors within 1 week prior to first dose of ModraDoc006/r. Single dose palliative radiation for pain relieve is allowed until one week prior to start with ModraDoc006/r (these lesions are not to be included as target lesions)
2. Any treatment with investigational drugs (or investigational device) within 21 days prior to receiving the first dose of ModraDoc006/r
3. Previous treatment with a taxane for recurrent or metastatic breast cancer
4. Major surgical procedures within 21 days prior to providing informed consent
5. Active acute or chronic infection, which is not controlled by appropriate medication (at the discretion of the treating physician)
6. Uncontrolled or significant cardiovascular disease defined as New York Heart Association Classification III or IV
7. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the Investigator would impair study compliance
8. Any medical condition that in the opinion of the Investigator would contra-indicate or preclude participation within the clinical trial, or would put the patient at high risk for treatment-related complications
9. Previous malignancies within the last three years other than breast carcinoma, except successfully treated squamous/basal cell carcinoma of the skin, superficial bladder cancer, and in situ carcinoma of the cervix
10. Patients with symptomatic brain metastases. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anticonvulsant therapy for at least 6 weeks are allowed to enrol. Radiotherapy for brain metastasis must have been completed at least 6 weeks prior to start of study treatment. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT completed at screening, demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive anti-epileptic drugs or corticosteroid treatment indicated for brain metastasis
11. Patients with confirmed leptomeningeal metastases
12. Women who are pregnant or breast feeding
13. Known positivity for Human Immunodeficiency Virus HIV-1 or HIV-2 type
14. Patients with known active infection of hepatitis B, C, or E (patients who are anti-HBC positive but HBsAg negative are eligible to participate in this study)
15. Bowel obstructions or motility disorders that may influence the resorption of drugs as judged by the Investigator
16. Patients with unstable ascites, defined as need for palliative paracentesis or presence of a permanent peritoneal drain in the past 4 weeks prior to first dose of ModraDoc006/r. Enrolment in patients with peritonitis carcinomatosa and malignant ascites is allowed if there is no clinical and/or radiological known or suspected motility disorder within the 4 weeks prior to the first dose of ModraDoc006/r
17. Concomitant use of MDR, MRP, OATP1B1, OATP1B3 and CYP3A modulating drugs such as Ca+- entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, and grapefruit juice, concomitant use of HIV medications, other protease inhibitors, (non) nucleoside analogues, or St. John's wort (see section 5.8). These need to have been stopped at least 5 times the terminal half-life (according to Summary of Product Characteristics (SPC)) or 7 days, whichever is longest, in order to prevent interaction with the drug. Tamoxifen and megestrol need to be stopped only 1 week prior to start of the first dose of ModraDoc006/r
18. Legal incapacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) | From baseline through study completion, an average of 1 year
  Evaluation of objective response rate that will be observed as measured by RECIST v1.1 criteria, in patients with recurrent or metastatic HER2 negative breast cancer after treatment with ModraDoc006/r

SECONDARY OUTCOMES:
The number of CTCAE v.4.03 toxicities during treatment with ModraDoc006/r | Evaluation of toxicities during the complete study treatment until 28 days after the last intake, using the CTCAEv4.03 grading system
  The hematological and non-hematological toxicity profile of ModraDoc006/r will be assessed by clinical and lab evaluation and evaluated according to CTCAE v.4.03
The activity data on progression-free survival (PFS) of ModraDoc006/r | From baseline through study completion, an average of 1 year
  Evaluation of progression free interval (PFS) that will be observed as measured by RECIST v1.1 criteria, in patients with recurrent or metastatic HER2 negative breast cancer during and after treatment with ModraDoc006/r

OTHER OUTCOMES:
The number of CTCAE v.4.03 toxicities during treatment with ModraDoc006/r in a population of frail patients | Evaluation of toxicities during the complete study treatment until 28 days after the last intake, using the CTCAEv4.03 grading system
  The hematological and non-hematological toxicity profile of ModraDoc006/r in frail patients will be assessed by clinical and lab evaluation and evaluated according to CTCAE v.4.03

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Keessen, Study Director — Modra Pharmaceuticals
Locations (4):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Universitaire de Liège, Liège
- Odense University Hospital, Odense, Denmark
- Hospital Quiron Pozuelo, Madrid, Spain